CLINICAL TRIAL: NCT01747096
Title: Diagnostic, Prospective, Comparative, Multicentric Study of the PET / CT With 68Ga-DOTANOC Versus Conventional Imaging Procedures (octréoscan ® Scintigraphy and CT / MRI) in the Assessment of in Gastroenteropancreatic Neuroendocrine Tumors
Brief Title: TEP With 68-DOTANOC in Gastroenteropancreatic Neuroendocrine Tumors
Acronym: 68-DOTANOC-GEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BRD/11/05-K
Record Dates: First submitted 2012-11-13; First posted 2012-12-11 (Estimated); Last update posted 2022-01-21 (Actual); Status verified 2016-07

CONDITIONS: Patients With Gastroenteropancreatic Neuroendocrine Tumors
Keywords: Gastroenteropancreatic Neuroendocrine Tumors; immuno PET (iPET); Gallium (68-Ga); DOTANOC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 68-Ga-DOTANOC (Experimental)
  Interventions: Drug: 68-Ga-DOTANOC

INTERVENTIONS:
Drug: 68-Ga-DOTANOC

SUMMARY:
Evaluation of the diagnostic performance of PET / CT with 68Ga-DOTANOC in Gastroenteropancreatic Neuroendocrine Tumors with comparison with other techniques used in routine clinical practice (octreoscan ® ; multiphase SPECT / CT, MRI or endoscopy).

Therapeutic impact and safety of PET / CT with 68Ga-DOTANOC will also be assessed. Expected results are a confirmation of the superiority of 68Ga-PET DOTANOC versus scintigraphy octreoscan ®, with a potential impact on the therapeutic management of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* effective contraception or exclusion of pregnancy dosage of beta-HCG in women of childbearing age
* Fortuitous discovery of suggestive tumors of TE-GEP with well documented conventional imaging (multiphase CT; MRI, US endoscopy) associated or not associated with clinical or biological signs of TE-GEP tumors (increase in tumor markers) OR
* Histologically proven GEP-TE (WHO classification 2010 (26) well differentiated in the initial staging OR
* Suspicion of recurrence or progression of well differentiated TE-GEP tumors on conventional imaging or laboratory tests (increase in tumor markers) OR
* Clinical or biological syndrome strongly suggestive of digestive endocrine disease without identification of lesions with conventional imaging
* Informed consent and patient's written
* Affiliation to an insurance

Exclusion Criteria:

* Multiple endocrine neoplasia
* TE GEP tumor not differentiated
* Pregnancy and lactation
* Persons protected by law
* Restlessness, inability to lie still hold at least 1 hour; Claustrophobia
* Poor compliance predictable or inability to undergo medical test for geographical, social or psychological
* Treatment with radiotherapy, chemotherapy or other antitumor treatment within 6 weeks of previous morphological and scintigraphic examinations. In case of treatment with somatostatin analogues delayed, scans will be performed 4 weeks after the last injection. However, a shorter period may be observed to avoid to do again the initial assessment exams.
* malignancy except basal cell cancers and cancer in situ of the cervix
* Contraindication of injection of a contrast agent necessary for the production of multiphase scanner.
* Patients who had a CT scan without injection of contrast material can not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Detection of Gastroenteropancreatic Neuroendocrine Tumors lesions in the initial assessment or during the search of recurrence. | 12 months
  Reference to the gold standard (that will be obtained from the data of histology and / or follow-up imaging at least 12 months

SECONDARY OUTCOMES:
Compare the diagnostic performance of PET / CT with 68Ga-DOTANOC with the standard process | 12 months

OTHER OUTCOMES:
Assess the clinical impact of PET / CT 68 Ga-DOTANOC in terms of specificity and predictive value for the detection of locations of GEP. | 12 months
Assess the relevance of decisions of PET / CT 68 Ga-DOTANOC in terms of specificity and predictive value for the detection of locations of GEP. | 12 months
Assess the value of PET / CT 68 Ga-DOTANOC in terms of specificity and predictive value for the detection of locations of GEP. | 12 months
Tolerance of 68-Ga-DOTANOC | 12 mois
  the vital signs and clinical tolerance will be assess during the 2 hours following injection of the radiopharmaceutical.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Ansquer, MD, Principal Investigator — Nantes Hospital
Locations (5):
- France (5):
  - Angers Hospital, Angers
  - Hôpital Beaujon, Clichy
  - Hôpital Bichat, Paris
  - Institut de Cancérologie de l'Ouest, René Gauducheau, Saint-Herblain
  - Nantes Hospital, Saint-Herblain